CLINICAL TRIAL: NCT04594876
Title: Cervical Epidural Versus Cevical Facet Injection for Patients With Chronic Cervical Pain
Acronym: D228
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Principal investigator, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D228; D228 (Registry Identifier: Faculty of medicine ethical committee, Fayoum university)
Record Dates: First submitted 2020-09-07; First posted 2020-10-20 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Intervention; Cervical; Epidural; Injection
Keywords: Flouroscopy; Cervical epidural; Facet injection; Neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Group P will receive cervical epidural Group F will receive cervical facet injection Both under fluroscopic guidance
Who Masked: Investigator
Masking Description: The patients were randomly allocated by a computer-generated table into one of two study groups. The randomization sequence was concealed in opaque sealed envelopes. The envelopes were opened by the study investigators just after recruitments and admission to the operation room. Only assessors and data collectors were blinded to the group's allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flouroscopic guidance Cervical Epidural injection (Other): Group (P) flouroscopic guidance cervical epidural injection
  Interventions: Other: Flouroscopic guidance cervical epidural versus cervical facet injection
- Flouroscopic guidance cervical facet injection (Other): Group (F) Flouroscopic guidance cervical facet injection
  Interventions: Other: Flouroscopic guidance cervical epidural versus cervical facet injection

INTERVENTIONS:
Other: Flouroscopic guidance cervical epidural versus cervical facet injection — The patients are classified in two groups group P for cervical epidural and group F for facet injection. The skin will be prepared with an antiseptic solution. The midline of the selected interspace will be identified under fluroscopic guidance.

SUMMARY:
After approval of the institutional review board and the Ethics Committee of Al Fayoum University number (D228) , and written informed consent from all patientṣ Pilot study will be done to confirm this sample size .The patients are classified in two groups group P for cervical epidural and group F for facet injection To compare effectivness of cervical epidural versus cervical facet injection under fluroscopic guidance in patients sufferring from chronic neck pain.

DETAILED DESCRIPTION:
After the approval of the institutional review board and the Ethics Committee of Al Fayoum University number (D228) , and written informed consent from all patientṣ Pilot study will be done to confirm this sample size .The patients are classified in two groups group P for cervical epidural and group F for facet injection. Patients Inclusion criteria of chronic cervical pain syndromes will be made from their history, symptoms, and imaging diagnosis. Patients will be lying down on the prone position. In group( F) Under the C-arm fluoroscopic guidance targeted zygapophyseal joints will be identified. The mixture of 2 mL of 2% lidocaine with 2 ml of beta methasone (6 mg/ml) will be injected in the joints unilaterally or bilaterally according to complaints of patients. Another group ( P) patients will undergo translaminar or interspinous cervical epidural block (CEBs). The translaminar or interlaminar approach is considered the safest and most effective technique for cervical epidural placement.The patient will be in a prone position. This procedure will be performed with fluoroscopic guidance. The patient will be placed in an optimal flexed cervical spine posture stabilized with enough resistance to prevent movement of the head during the procedure. The skin will be prepared with an antiseptic solution. The midline of the selected interspace will be identified under fluroscopic guidance. LA, such as lidocaine, will be used, to mark the intended site of skin entry. As much as 1 mL of lidocaine will be used to infiltrate the skin and subcutaneous tissues. We will insert a 25-gauge, 2-inch needle exactly into the targeted midline. After the LA has been given time to anesthetize the area,we will hold the needle firmly at the hub with the left thumb and index finger. Then the palm of the left hand will be placed firmly against the patient's neck, so that the left hand acts as a unit to stabilize, protect, and control the needle's trajectory and its metered ingress from any unexpected patient activity. The needle will be then advanced with the left hand, which is braced against the neck with the needle hub held tightly between the left thumb and forefinger. We will use the right hand to monitor resistance through a syringe containing air. With constant pressure applied to the plunger of the syringe through light pressure applied by the right thumb, the needle and syringe will be advanced in a slow and deliberate manner. As the bevel passes through the ligament flavum and enters the epidural space, a sudden loss of resistance that we will appreciate also we can appreciate the entrence the epidural space under fluroscopic guidance in condition that not to cross J line (a line appear under flouroscopy imaging facet joint articulation if crossing this line we will puncture the dura).

Needle position within the epidural space will be checked by using fluoroscopic verification and by repeating the loss of resistance maneuver. The cervical epidural space should accept 0.5-1 mL of air or sterile preservative free saline without significant resistance. The force required to depress the plunger should not exceed that which is necessary to overcome the resistance of the needle. Any significant pain or sudden increase in resistance during the injection suggests incorrect needle placement, so the injection will be stopped and we will assess the position of the needle using fluoroscopy. If the needle remains satisfactorily placed and loss of resistance within the epidural space is confirmed without additional patient report of pain, gentle aspiration will be checked to assure that the needle is not positioned in the subarachnoid space or that it's not intravascular. If cerebrospinal fluid (CSF) is aspirated, we will repeat the block attempt at a different interspace. If aspiration of blood occurs, the needle will be tightly rotated and the aspiration test will be repeated. If the aspiration of blood continues, the procedure will be aborted due to the danger of developing an epidural hematoma and possibly neurological compromise. when the needle is correctly placed in the midline of the epidural space, then injection of the mixture of 2 mL of 2% lidocaine with 2 ml of beta methasone (6 mg/ml) will be done .

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20 - 70 years old.
* ASA I and II
* Cervical pain at least 3 months before procedure
* Patients have failed pharmacological treatment.

Exclusion Criteria:

* Systemic infection
* Skin infection
* Bleeding tendency and coagulopathy
* Pregnancy
* Neurological disorders
* Any deformaties that disfacilate the procedure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Neck pain disability index preintervention | measured once within 1 day pre intervention
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain and is used by clinicians and researchers alike.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score. Occasionally, a respondent will not complete one question or another. The average of all other items is then added to the completed items.
  The original report provided scoring intervals for interpretation, as follows:
  0 - 4 = no disability 5 - 14 = mild 15 - 24 = moderate 25 - 34 = severe above 34 = complete.
Change in Neck pain disability index post intervention | 1 month, 3 month, 6 month,12 month
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain and is used by clinicians and researchers alike.
  Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score. Occasionally, a respondent will not complete one question or another. The average of all other items is then added to the completed items.
  The original report provided scoring intervals for interpretation, as follows:
  0 - 4 = no disability 5 - 14 = mild 15 - 24 = moderate 25 - 34 = severe above 34 = complete.

OTHER OUTCOMES:
Total opoid and non steroidal consumption preintervention | measured once 1 day preintervention
  Pre intervention total dose of opoid and an non steroid consumption
Total opoid and non steroidal consumption post intervention | measured (1 month,3 month,6 month,12 month)"post intervention
  Total dose intake of opoid and non steroid consumption post intervention
VAS Score | 0 hour, 2 hours, 4 hours, 6hours, 12 hours, 18 hours, 24 hours post operative
  Graded frome 0 no pain to 10 maximum pain
Post operative Nausea & vomiting score | 0 hour,2 hours,4 hours,6 hours,12 hours,18 hours,24 hours post operative
  From grade 0 no nausea or vomiting to grade 4 sever vomitting

CONTACTS AND LOCATIONS:
Overall Officials: Atef Mahmoud, Principal Investigator — Fayoum University Hospital
Locations (1):
- Atef Mohamed mahmoud, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No
The study will be start after completion It will available